CLINICAL TRIAL: NCT05475808
Title: Comparison of the Efficacy of Different Treatment Methods in Patients With Carpal Tunnel Syndrome
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-SK-02
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Splint (Active Comparator): Patients in Group 1 will be applied to only static wrist splint treatment for 8 week.
  Interventions: Device: Static wrist splint treatment
- Tendon and nerve gliding exercise (Active Comparator): Patients in Group 2 will be applied to tendon and nerve gliding exercises for the wrist in addition to static wrist splint treatment for 8 week.
  Interventions: Device: Static wrist splint treatment; Other: Tendon and nerve gliding exercises
- local steroid injection (Active Comparator): Patients in Group 3 will be applied to local steroid injection to wrist in addition to static wrist splint treatment for 8 week.
  Interventions: Device: Static wrist splint treatment; Drug: Wrist local steroid injection

INTERVENTIONS:
Device: Static wrist splint treatment — Static wrist splint (volar wrist cock-up orthosis): It extends from the proximal of the metacarpophalangeal (MCP) joint to the distal 2/3 of the forearm, supports the wrist from the volar face. It stabilizes the wrist in 20-30 degrees of dorsiflexion and restricts wrist movements. It allows movement of the MCP joints. Patients will be asked to wear this splint continuously at night and for at least 4 hours during the day for 8 weeks.
Other: Tendon and nerve gliding exercises — Tendon and nerve gliding exercises will be applied 5 sessions a day for 8 weeks. Each session will hold 10 repetitions and approximately 7 seconds in each exercise position.
  These exercises involve a sequence of finger movements (for tendon gliding) and wrist and fingers movements (for median nerve gliding).
  Arms: Tendon and nerve gliding exercise
Drug: Wrist local steroid injection — Wrist local steroid injection:
  After proper area cleaning with povidone solution, 1ml Betamethasone dipropionate + Betamethasone sodium phosphate (6.43 mg/ml + 2.63 mg/ml) steroid injection will be applied around the median nerve with a 22 G injector from ulnar side of the wrist proximal crease under ultrasound guidance.
  Arms: local steroid injection

SUMMARY:
It is aimed to compare the effects of different conservative methods on the clinical condition of the patients, hand grip and pinch strengths and wrist muscle strengths in patients with carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is one of the most common entrapment neuropathies. It occurs as a result of compression or irritation of the median nerve as it passes through the carpal tunnel in the wrist. It is seen in 1-4% of the general population.In nerve conduction studies, patients with mild and moderate CTS are treated with conservative treatment methods, while patients with severe nerve conduction findings and thenar atrophy are treated surgically.Although there are many methods used in the conservative treatment of carpal tunnel syndrome, there is no definite data about which treatment option to choose.The most commonly used conservative method is the wrist rest splint application, which is based on the principle of resting the wrist.In addition, there are tendon and nerve gliding exercises that facilitate nerve and tendon movements. Physical therapy agents such as Tens, Laser and Ultrasound can be used in the treatment of CTS. Non-Steroidal anti-inflammatory drugs and B6 vitamins can be used as drug therapy. Apart from these, local corticosteroid injections can be applied from the wrist.

There are studies comparing conservative treatment methods in carpal tunnel syndrome. However, these are generally in the form of studies that measure and compare the effects of treatments on the clinical condition of their patients and on hand grip and finger pinch strength. There is no comparative study investigating the effects of conservative treatment methods on wrist muscle strength in patients with carpal tunnel syndrome.

It was observed that wrist muscle strength decreased in patients with CTS compared to normal patients. Wrist muscle strength is important in hand and wrist functions as well as hand grip and pinch strength are important.

Flexion-extension, radial-ulnar deviation and supination-pronation muscle strengths of the patients' wrists can be measured with an isokinetic dynamometer device.

It is aimed to compare the effects of different conservative methods on the clinical condition of the patients, hand grip and pinch strengths and wrist muscle strengths in patients with carpal tunnel syndrome.

It will be organized as a prospective randomized study. It is planned to include 60 patients in the study. Patients will be randomized into three groups in equal numbers, stratified by age and sex.

Patients in Group 1 will be applied to only static wrist splint treatment for 8 week.

Patients in Group 2 will be applied to tendon and nerve gliding exercises for the wrist in addition to static wrist splint treatment for 8 week .

Patients in Group 3 will be applied to local steroid injection the wrist in addition to static wrist splint treatment for 8 week.

Demographic data, medical history, dominant and CTS hand information will be recorded at the beginning of the patients.

Patients in both groups will be evaluated before the treatment, at the 8th week after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate CTS confirmed by Electromyography
* Clinically, at least one of the symptoms of hand-wrist pain, numbness, night pain should be present.
* Clinically, at least one of the Tinel, Phalen, and median nerve compression findings should be present.

Exclusion Criteria:

* Having a history of trauma and operation on the wrist.
* Patients who have had previous injections from the wrist
* Patients with thyroid diseases, diabetes mellitus, systemic peripheral neuropathy and cervical radiculopathy
* Pregnant patients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2025-05-27 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Before Treatment
  Pain was evaluated using a 10 cm long Visual Analogue Scale (VAS) during rest and activity (0 = no pain, 10 = very severe pain).
Visual Analogue Scale | 8 week after treatment
  Pain was evaluated using a 10 cm long Visual Analogue Scale (VAS) during rest and activity (0 = no pain, 10 = very severe pain).
Isokinetic Muscle Strength Measure | Before Treatment
  Wrist flexion/extension, radial/ulnar deviation, supination/pronation strengths at 60° and 210°/s will be evaluated with an isokinetic test and exercise system (CSMI Cybex). Patients will be seated on the test chair with the backrest set to 90°. The arm to be tested will be secured to the chair's forearm rest. The wrist joint will be positioned in neutral. The forearm stabilizer pad and strap will secure the distal aspect of the forearm of the test hand. Wrist flexion/extension range of motion, radial/ulnar deviation range of motion, supination/pronation range of motion will be set within each patients' available range. Patients will be permitted 4 experimental trials to become familiar with the process for each angular velocity, and then they will perform 5 maximal repetitions at 60°/s and 12 maximal repetitions at 210°/s. At the end of the test, muscle strength (Peak Torque) will be measured in Newton meters.
Isokinetic Muscle Strength Measure | 8 week after treatment
  Wrist flexion/extension, radial/ulnar deviation, supination/pronation strengths at 60° and 210°/s will be evaluated with an isokinetic test and exercise system (CSMI Cybex). Patients will be seated on the test chair with the backrest set to 90°. The arm to be tested will be secured to the chair's forearm rest. The wrist joint will be positioned in neutral. The forearm stabilizer pad and strap will secure the distal aspect of the forearm of the test hand. Wrist flexion/extension range of motion, radial/ulnar deviation range of motion, supination/pronation range of motion will be set within each patients' available range. Patients will be permitted 4 experimental trials to become familiar with the process for each angular velocity, and then they will perform 5 maximal repetitions at 60°/s and 12 maximal repetitions at 210°/s. At the end of the test, muscle strength (Peak Torque) will be measured in Newton meters.
The hand grip strength | Before Treatment
  The hand grip strength of the patients will be measured with a North Coast hydraulic hand dynamometer. The average of 3 different repetitive measurements will be taken.
The hand grip strength | 8 week after treatment
  The hand grip strength of the patients will be measured with a North Coast hydraulic hand dynamometer. The average of 3 different repetitive measurements will be taken.
The finger pinch strength | Before Treatment
  Finger pinch strength will be measured with a North Coast hydraulic pinch gauge. The average of 3 different repetitive measurements will be taken.
The finger pinch strength | 8 week after treatment
  Finger pinch strength will be measured with a North Coast hydraulic pinch gauge. The average of 3 different repetitive measurements will be taken.
Boston Carpal Tunnel Syndrome Questionnaire | Before Treatment
  This questionnaire consists of two parts: Boston Symptom Severity Scale (BSSS) and Boston Functional Capacity Scale (BFCS). BSSS consists of 11 questions, and BFCS consists of 8 questions. The score of each question varies between 1-5. High scores indicate severe symptoms and reduced functional capacity.
Boston Carpal Tunnel Syndrome Questionnaire | 8 week after treatment
  This questionnaire consists of two parts: Boston Symptom Severity Scale (BSSS) and Boston Functional Capacity Scale (BFCS). BSSS consists of 11 questions, and BFCS consists of 8 questions. The score of each question varies between 1-5. High scores indicate severe symptoms and reduced functional capacity.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder end Hand Questionnaire | Before Treatment
  The Disabilities of the Arm, Shoulder end Hand Questionnaire (DASH) consists of 3 parts: the functional/symptom model, the business model, and the sports/musicians model. The individual fills himself. In this study, functional/symptom and business model sections will be used. A score between 0-100 is obtained from each section. High score increases handicap.
Disabilities of the Arm, Shoulder end Hand Questionnaire | 8 week after treatment
  The Disabilities of the Arm, Shoulder end Hand Questionnaire (DASH) consists of 3 parts: the functional/symptom model, the business model, and the sports/musicians model. The individual fills himself. In this study, functional/symptom and business model sections will be used. A score between 0-100 is obtained from each section. High score increases handicap.
Short Form-36 Quality of Life Scale | Before Treatment
  The patients' quality of life will be evaluated with the Short Form-36 Quality of Life Scale. It consists of 36 questions filled by the individual himself. High scores indicate good quality of life.
Short Form-36 Quality of Life Scale | 8 week after treatment
  The patients' quality of life will be evaluated with the Short Form-36 Quality of Life Scale. It consists of 36 questions filled by the individual himself. High scores indicate good quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)